CLINICAL TRIAL: NCT00591357
Title: Study of the Efficacy of Loperamide in Treating Patients for Clostridium Difficile Colitis and Diarrheal Disease of Unknown Cause Associated With Prior Antibiotic Therapy.
Brief Title: Efficacy of Loperamide for C. Difficile Colitis and Other Diarrheal Diseases Associated With Antibiotic Therapy
Acronym: loperamide
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of personnel to complete trial
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Daniel M. Musher MD, Principal Investigator, Michael E. DeBakey VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-21387; Clostridium difficile; Antibiotic associated diarrhea; loperamide
Record Dates: First submitted 2007-12-31; First posted 2008-01-11 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Antibiotic-Associated Diarrhea; Clostridium Difficile
Keywords: Antibiotic associated diarrhea; Clostridium difficile; loperamide
MeSH Terms: interventions — Loperamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Loperamide
  Interventions: Drug: loperamide
- B (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: loperamide — 4 mg PO initially and 2 mg after each water stoll not to exceed 10 mg qd
  Arms: A
Drug: placebo — 4 mg PO initially and 2 mg after each water stoll not to exceed 10 mg qd
  Arms: B

SUMMARY:
To determine whether symptomatic treatment of the diarrhea in CDAD reduces morbidity and mortality of this serious nosocomial infection in patients who have antibiotic-associated diarrhea. Both C. diff positive and negative patients will be included.

DETAILED DESCRIPTION:
Colitis due to Clostridium difficile has been increasingly recognized as a serious nosocomial problem. Recommended therapy is with metronidazole, 500 mg four times daily for 10 days. About 80% of patients respond to this therapy. However, the response may be be delayed, in which case debilitation due to diarrhea progresses. The 20% who do not respond tend to be sicker to start, and debilitation due to diarrhea is a severe problem. In reviewing the medical literature, we discovered that the earliest papers on C. difficile colitis emphasized symptomatic therapy with 'lomotil' (diphenoxylate with atropine).

Treatment to suppress the diarrhea fell out of favor in the late 1970's because of the theoretical consideration that it was better to expel than to retain the bacterial toxins. However, the patients who are affected by C. difficile colitis are increasingly elderly and debilitated, and suffer substantial morbidity from the diarrhea. We have shown that the 90-day associated mortality is >20%.

Loperamide is a standard treatment for diarrhea, and is available over the counter under the name, Imodium. Based on a few anecdotal reports, this drug is regarded as contraindicated in patients whose diarrheal disease is bacterial. But it is used widely, and generally without any diagnosis being established. We now propose to administer loperamide or placebo to patients with CDAD in order to determine whether the antidiarrheal drug reduces morbidity associated with the infection. We will monitor our patients closely both to observe potential benefits and/or adverse events.

In the addendum, we propose to include patients who have antibiotic-associated diarrheal disease that is not due to C. difficile. There are many patients who have antibiotic-associated diarrheal disease who test negative for C. difficile. We believe that these patient may benefit from loperamide treatment as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diarrheal stools considered to be antibiotic associated

Exclusion Criteria:

* Inability of sign consent
* Patient with other known gastrointestinal disease
* Patients receiving tube feeding or fecal incontinence prior to receiving antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-10; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To determin symptomatic treatment of diarrhea with loperamide in antibiotic associated diarrhea | 2 years

SECONDARY OUTCOMES:
To measure the safety and efficacy of loperamide in the control of antibiotic associated diarrhea in hospitalized patients | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Musher, MD, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- VAMC, Houston, Texas, United States